CLINICAL TRIAL: NCT03220776
Title: Imaging Framework for Testing GABAergic/Glutamatergic Drugs in Bipolar Alcoholics
Brief Title: Imaging GABAergic/Glutamatergic Drugs in Bipolar Alcoholics Alcoholics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, James J. Prisciandaro, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 64964; R01AA025365 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Alcohol Use Disorder; Bipolar Disorder
MeSH Terms: conditions — Alcoholism; Bipolar Disorder | interventions — Acetylcysteine; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Gabapentin, then N-Acetylcysteine, then Placebo Oral Capsule (Experimental): Three, 1-week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Interventions: Drug: N-Acetylcysteine; Drug: Gabapentin; Drug: Placebo Oral Tablet
- N-Acetylcysteine, then Placebo Oral Capsule, then Gabapentin (Experimental): 3, 1 week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Interventions: Drug: N-Acetylcysteine; Drug: Gabapentin; Drug: Placebo Oral Tablet
- Placebo Oral Tablet, then Gabapentin, then N-Acetylcysteine (Placebo Comparator): Three, 1-week conditions. Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Interventions: Drug: N-Acetylcysteine; Drug: Gabapentin; Drug: Placebo Oral Tablet
- Placebo Oral Capsule, then N-Acetylcysteine, then Gabapentin (Experimental): Three, 1-week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Interventions: Drug: N-Acetylcysteine; Drug: Gabapentin; Drug: Placebo Oral Tablet
- Gabapentin, then Placebo Oral Capsule, then N-Acetylcysteine (Experimental): Three, 1-week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Interventions: Drug: N-Acetylcysteine; Drug: Gabapentin; Drug: Placebo Oral Tablet
- N-Acetylcysteine, then Gabapentin, then Placebo Oral Capsule (Experimental): Three, 1-week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Interventions: Drug: N-Acetylcysteine; Drug: Gabapentin; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: N-Acetylcysteine — 5 day trial of N-acetylcysteine with titration to 2,400mg
Drug: Gabapentin — 5 day trial of gabapentin with titration to 1,200mg
Drug: Placebo Oral Tablet — 5 day trial of matched placebo

SUMMARY:
The proposed 3-week, double-blind, crossover, proof of concept study aims to manipulate neurochemical dysfunctions characteristic of individuals with co-occurring BD and AUD (i.e., abnormally low prefrontal GABA and glutamate), using medications that have been shown to normalize cortical GABA (i.e., gabapentin) and glutamate (i.e., NAC) levels in past research, and to evaluate medication-related changes in response inhibition and alcohol cue-reactivity fMRI tasks as well as drinking and mood in individuals with AUD+BD.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is the Axis I psychiatric condition most strongly associated with substance use disorder (SUD); diagnostic co-occurrence is particularly high between BD and alcohol use disorder (AUD). Individuals with co-occurring SUD and BD (SUD+BD) have substantially worse clinical outcomes than those with either BD or SUD alone. Nonetheless, little is known about optimal treatment for individuals with SUD+BD; response to lithium appears to be poor, and only one double-blind, randomized, placebo-controlled trial of valproate has demonstrated improved drinking outcomes in this population. Traditionally, treatment trials for SUD+BD have investigated medications that have been FDA approved to treat either BD or SUD in hopes that such medications would prove efficacious in individuals with SUD+BD. A different approach to selecting, and ideally developing, medications for SUD+BD treatment trials would be to target neurochemical dysfunctions characteristic of individuals with both BD and SUD. Recent research by the current investigator has demonstrated unique disturbances in prefrontal gamma-Aminobutyric acid (GABA) and glutamate concentrations in this population using proton magnetic resonance spectroscopy (1H-MRS), with individuals with co-occurring alcohol dependence (AD) and BD having significantly lower levels of GABA and glutamate relative to individuals with BD alone, AD alone, or healthy controls. Lower levels of prefrontal GABA and glutamate were in turn associated with elevated impulsivity and alcohol craving. The proposed 3-week, double-blind, crossover, proof of concept study will evaluate: a) whether medications that have been demonstrated to normalize cortical GABA (i.e., gabapentin) and glutamate (i.e., N-Acetylcysteine [NAC]) concentrations in individuals with epilepsy and cocaine dependence, respectively, may similarly act to normalize prefrontal GABA and glutamate levels in individuals with AUD+BD, and b) whether normalization of prefrontal GABA and glutamate levels will be associated with improvements in functional brain activity to tasks that assess core neurobehavioral deficits of AUD and BD (i.e., response inhibition, alcohol cue-reactivity), as well as drinking and mood symptoms. Positive results may support investigation of gabapentin and/or NAC as adjunctive treatments for AUD+BD in large-scale, randomized clinical trials. Most importantly, the proposed study may provide successful demonstration of a neuro-behavioral, multimodal neuroimaging platform for evaluating the potential promise of GABAergic and glutamatergic drugs for AUD and/or BD, as well as other conditions marked by GABAergic/glutamatergic dysfunction.

ELIGIBILITY:
Inclusion:

* Meets DSM-V diagnostic criteria for Bipolar Disorder
* Using at least one mood stabilizing medication
* Meets diagnostic criteria Alcohol Use Disorder, with active drinking in the past month.

Exclusion:

* Serious medical or non-inclusionary psychiatric disease
* Concomitant use of benzodiazepine medications or any medications hazardous if taken with gabapentin/N-acetylcysteine
* History of clinically significant brain injury
* Presence of non-MRI safe material, or clinically significant claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J Prisciandarao, Ph. D, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altshuler LL, Bookheimer SY, Townsend J, Proenza MA, Eisenberger N, Sabb F, Mintz J, Cohen MS. Blunted activation in orbitofrontal cortex during mania: a functional magnetic resonance imaging study. Biol Psychiatry. 2005 Nov 15;58(10):763-9. doi: 10.1016/j.biopsych.2005.09.012. PMID 16310510
- [Background] Anton RF, Moak DH, Latham P. The Obsessive Compulsive Drinking Scale: a self-rated instrument for the quantification of thoughts about alcohol and drinking behavior. Alcohol Clin Exp Res. 1995 Feb;19(1):92-9. doi: 10.1111/j.1530-0277.1995.tb01475.x. PMID 7771669
- [Background] Anton RF, Myrick H, Baros AM, Latham PK, Randall PK, Wright TM, Stewart SH, Waid R, Malcolm R. Efficacy of a combination of flumazenil and gabapentin in the treatment of alcohol dependence: relationship to alcohol withdrawal symptoms. J Clin Psychopharmacol. 2009 Aug;29(4):334-42. doi: 10.1097/JCP.0b013e3181aba6a4. PMID 19593171
- [Background] Anton RF, Myrick H, Wright TM, Latham PK, Baros AM, Waid LR, Randall PK. Gabapentin combined with naltrexone for the treatment of alcohol dependence. Am J Psychiatry. 2011 Jul;168(7):709-17. doi: 10.1176/appi.ajp.2011.10101436. Epub 2011 Mar 31. PMID 21454917
- [Background] Aufhaus E, Weber-Fahr W, Sack M, Tunc-Skarka N, Oberthuer G, Hoerst M, Meyer-Lindenberg A, Boettcher U, Ende G. Absence of changes in GABA concentrations with age and gender in the human anterior cingulate cortex: a MEGA-PRESS study with symmetric editing pulse frequencies for macromolecule suppression. Magn Reson Med. 2013 Feb;69(2):317-20. doi: 10.1002/mrm.24257. Epub 2012 Apr 5. PMID 22488982
- [Background] Bagga D, Khushu S, Modi S, Kaur P, Bhattacharya D, Garg ML, Singh N. Impaired visual information processing in alcohol-dependent subjects: a proton magnetic resonance spectroscopy study of the primary visual cortex. J Stud Alcohol Drugs. 2014 Sep;75(5):817-26. doi: 10.15288/jsad.2014.75.817. PMID 25208200
- [Background] Bak LK, Schousboe A, Waagepetersen HS. The glutamate/GABA-glutamine cycle: aspects of transport, neurotransmitter homeostasis and ammonia transfer. J Neurochem. 2006 Aug;98(3):641-53. doi: 10.1111/j.1471-4159.2006.03913.x. Epub 2006 Jun 19. PMID 16787421
- [Background] Baker DA, McFarland K, Lake RW, Shen H, Tang XC, Toda S, Kalivas PW. Neuroadaptations in cystine-glutamate exchange underlie cocaine relapse. Nat Neurosci. 2003 Jul;6(7):743-9. doi: 10.1038/nn1069. PMID 12778052
- [Background] Bauer J, Pedersen A, Scherbaum N, Bening J, Patschke J, Kugel H, Heindel W, Arolt V, Ohrmann P. Craving in alcohol-dependent patients after detoxification is related to glutamatergic dysfunction in the nucleus accumbens and the anterior cingulate cortex. Neuropsychopharmacology. 2013 Jul;38(8):1401-8. doi: 10.1038/npp.2013.45. Epub 2013 Feb 12. PMID 23403696
- [Background] Beck A, Schlagenhauf F, Wustenberg T, Hein J, Kienast T, Kahnt T, Schmack K, Hagele C, Knutson B, Heinz A, Wrase J. Ventral striatal activation during reward anticipation correlates with impulsivity in alcoholics. Biol Psychiatry. 2009 Oct 15;66(8):734-42. doi: 10.1016/j.biopsych.2009.04.035. Epub 2009 Jun 27. PMID 19560123
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Behar KL, Rothman DL, Petersen KF, Hooten M, Delaney R, Petroff OA, Shulman GI, Navarro V, Petrakis IL, Charney DS, Krystal JH. Preliminary evidence of low cortical GABA levels in localized 1H-MR spectra of alcohol-dependent and hepatic encephalopathy patients. Am J Psychiatry. 1999 Jun;156(6):952-4. doi: 10.1176/ajp.156.6.952. PMID 10360140
- [Background] Benes FM, Berretta S. GABAergic interneurons: implications for understanding schizophrenia and bipolar disorder. Neuropsychopharmacology. 2001 Jul;25(1):1-27. doi: 10.1016/S0893-133X(01)00225-1. PMID 11377916
- [Background] Berk M, Copolov DL, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Bush AI. N-acetyl cysteine for depressive symptoms in bipolar disorder--a double-blind randomized placebo-controlled trial. Biol Psychiatry. 2008 Sep 15;64(6):468-75. doi: 10.1016/j.biopsych.2008.04.022. Epub 2008 Jun 5. PMID 18534556
- [Background] Berk M, Dean O, Cotton SM, Gama CS, Kapczinski F, Fernandes BS, Kohlmann K, Jeavons S, Hewitt K, Allwang C, Cobb H, Bush AI, Schapkaitz I, Dodd S, Malhi GS. The efficacy of N-acetylcysteine as an adjunctive treatment in bipolar depression: an open label trial. J Affect Disord. 2011 Dec;135(1-3):389-94. doi: 10.1016/j.jad.2011.06.005. Epub 2011 Jun 29. PMID 21719110
- [Background] Bermpohl F, Kahnt T, Dalanay U, Hagele C, Sajonz B, Wegner T, Stoy M, Adli M, Kruger S, Wrase J, Strohle A, Bauer M, Heinz A. Altered representation of expected value in the orbitofrontal cortex in mania. Hum Brain Mapp. 2010 Jul;31(7):958-69. doi: 10.1002/hbm.20909. PMID 19950195
- [Background] Bhagwagar Z, Wylezinska M, Jezzard P, Evans J, Ashworth F, Sule A, Matthews PM, Cowen PJ. Reduction in occipital cortex gamma-aminobutyric acid concentrations in medication-free recovered unipolar depressed and bipolar subjects. Biol Psychiatry. 2007 Mar 15;61(6):806-12. doi: 10.1016/j.biopsych.2006.08.048. Epub 2007 Jan 8. PMID 17210135
- [Background] Bohn MJ, Krahn DD, Staehler BA. Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcohol Clin Exp Res. 1995 Jun;19(3):600-6. doi: 10.1111/j.1530-0277.1995.tb01554.x. PMID 7573780
- [Background] Boy F, Evans CJ, Edden RA, Lawrence AD, Singh KD, Husain M, Sumner P. Dorsolateral prefrontal gamma-aminobutyric acid in men predicts individual differences in rash impulsivity. Biol Psychiatry. 2011 Nov 1;70(9):866-72. doi: 10.1016/j.biopsych.2011.05.030. Epub 2011 Jul 14. PMID 21757187
- [Background] Brady RO Jr, McCarthy JM, Prescot AP, Jensen JE, Cooper AJ, Cohen BM, Renshaw PF, Ongur D. Brain gamma-aminobutyric acid (GABA) abnormalities in bipolar disorder. Bipolar Disord. 2013 Jun;15(4):434-9. doi: 10.1111/bdi.12074. Epub 2013 May 2. PMID 23634979
- [Background] Brennan BP, Hudson JI, Jensen JE, McCarthy J, Roberts JL, Prescot AP, Cohen BM, Pope HG Jr, Renshaw PF, Ongur D. Rapid enhancement of glutamatergic neurotransmission in bipolar depression following treatment with riluzole. Neuropsychopharmacology. 2010 Feb;35(3):834-46. doi: 10.1038/npp.2009.191. Epub 2009 Dec 2. PMID 19956089
- [Background] Brooks JO 3rd, Wang PW, Strong C, Sachs N, Hoblyn JC, Fenn R, Ketter TA. Preliminary evidence of differential relations between prefrontal cortex metabolism and sustained attention in depressed adults with bipolar disorder and healthy controls. Bipolar Disord. 2006 Jun;8(3):248-54. doi: 10.1111/j.1399-5618.2006.00310.x. PMID 16696826
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cai K, Nanga RP, Lamprou L, Schinstine C, Elliott M, Hariharan H, Reddy R, Epperson CN. The impact of gabapentin administration on brain GABA and glutamate concentrations: a 7T (1)H-MRS study. Neuropsychopharmacology. 2012 Dec;37(13):2764-71. doi: 10.1038/npp.2012.142. Epub 2012 Aug 8. PMID 22871916
- [Background] Carta MG, Hardoy MC, Hardoy MJ, Grunze H, Carpiniello B. The clinical use of gabapentin in bipolar spectrum disorders. J Affect Disord. 2003 Jun;75(1):83-91. doi: 10.1016/s0165-0327(02)00046-0. PMID 12781355
- [Background] Chang L, Jiang CS, Ernst T. Effects of age and sex on brain glutamate and other metabolites. Magn Reson Imaging. 2009 Jan;27(1):142-5. doi: 10.1016/j.mri.2008.06.002. Epub 2008 Aug 6. PMID 18687554
- [Background] Corr PJ. Reinforcement sensitivity theory and personality. Neurosci Biobehav Rev. 2004 May;28(3):317-32. doi: 10.1016/j.neubiorev.2004.01.005. PMID 15225974
- [Background] Dager SR, Friedman SD, Parow A, Demopulos C, Stoll AL, Lyoo IK, Dunner DL, Renshaw PF. Brain metabolic alterations in medication-free patients with bipolar disorder. Arch Gen Psychiatry. 2004 May;61(5):450-8. doi: 10.1001/archpsyc.61.5.450. PMID 15123489
- [Background] Edden RA, Puts NA, Harris AD, Barker PB, Evans CJ. Gannet: A batch-processing tool for the quantitative analysis of gamma-aminobutyric acid-edited MR spectroscopy spectra. J Magn Reson Imaging. 2014 Dec;40(6):1445-52. doi: 10.1002/jmri.24478. Epub 2013 Nov 13. PMID 25548816
- [Background] Ehrlich A, Schubert F, Pehrs C, Gallinat J. Alterations of cerebral glutamate in the euthymic state of patients with bipolar disorder. Psychiatry Res. 2015 Aug 30;233(2):73-80. doi: 10.1016/j.pscychresns.2015.05.010. Epub 2015 May 22. PMID 26050195
- [Background] Ende G, Cackowski S, Van Eijk J, Sack M, Demirakca T, Kleindienst N, Bohus M, Sobanski E, Krause-Utz A, Schmahl C. Impulsivity and Aggression in Female BPD and ADHD Patients: Association with ACC Glutamate and GABA Concentrations. Neuropsychopharmacology. 2016 Jan;41(2):410-8. doi: 10.1038/npp.2015.153. Epub 2015 Jun 4. PMID 26040503
- [Background] Ende G, Hermann D, Demirakca T, Hoerst M, Tunc-Skarka N, Weber-Fahr W, Wichert S, Rabinstein J, Frischknecht U, Mann K, Vollstadt-Klein S. Loss of control of alcohol use and severity of alcohol dependence in non-treatment-seeking heavy drinkers are related to lower glutamate in frontal white matter. Alcohol Clin Exp Res. 2013 Oct;37(10):1643-9. doi: 10.1111/acer.12149. Epub 2013 Jun 25. PMID 23800328
- [Background] Fatemi SH, Stary JM, Earle JA, Araghi-Niknam M, Eagan E. GABAergic dysfunction in schizophrenia and mood disorders as reflected by decreased levels of glutamic acid decarboxylase 65 and 67 kDa and Reelin proteins in cerebellum. Schizophr Res. 2005 Jan 1;72(2-3):109-22. doi: 10.1016/j.schres.2004.02.017. PMID 15560956
- [Background] Fazel S, Lichtenstein P, Grann M, Goodwin GM, Langstrom N. Bipolar disorder and violent crime: new evidence from population-based longitudinal studies and systematic review. Arch Gen Psychiatry. 2010 Sep;67(9):931-8. doi: 10.1001/archgenpsychiatry.2010.97. PMID 20819987
- [Background] Frye MA, Watzl J, Banakar S, O'Neill J, Mintz J, Davanzo P, Fischer J, Chirichigno JW, Ventura J, Elman S, Tsuang J, Walot I, Thomas MA. Increased anterior cingulate/medial prefrontal cortical glutamate and creatine in bipolar depression. Neuropsychopharmacology. 2007 Dec;32(12):2490-9. doi: 10.1038/sj.npp.1301387. Epub 2007 Apr 11. PMID 17429412
- [Background] Gass JT, Olive MF. Glutamatergic substrates of drug addiction and alcoholism. Biochem Pharmacol. 2008 Jan 1;75(1):218-65. doi: 10.1016/j.bcp.2007.06.039. Epub 2007 Jun 30. PMID 17706608
- [Background] Gerner RH, Fairbanks L, Anderson GM, Young JG, Scheinin M, Linnoila M, Hare TA, Shaywitz BA, Cohen DJ. CSF neurochemistry in depressed, manic, and schizophrenic patients compared with that of normal controls. Am J Psychiatry. 1984 Dec;141(12):1533-40. doi: 10.1176/ajp.141.12.1533. PMID 6209989
- [Background] Gibbons RD, Hur K, Brown CH, Mann JJ. Gabapentin and suicide attempts. Pharmacoepidemiol Drug Saf. 2010 Dec;19(12):1241-7. doi: 10.1002/pds.2036. Epub 2010 Oct 4. PMID 20922708
- [Background] Godlewska BR, Yip SW, Near J, Goodwin GM, Cowen PJ. Cortical glutathione levels in young people with bipolar disorder: a pilot study using magnetic resonance spectroscopy. Psychopharmacology (Berl). 2014 Jan;231(2):327-32. doi: 10.1007/s00213-013-3244-0. Epub 2013 Aug 17. PMID 23955702
- [Background] Goldberg JF, Garno JL, Leon AC, Kocsis JH, Portera L. A history of substance abuse complicates remission from acute mania in bipolar disorder. J Clin Psychiatry. 1999 Nov;60(11):733-40. doi: 10.4088/jcp.v60n1103. PMID 10584760
- [Background] Gomez R, Behar KL, Watzl J, Weinzimer SA, Gulanski B, Sanacora G, Koretski J, Guidone E, Jiang L, Petrakis IL, Pittman B, Krystal JH, Mason GF. Intravenous ethanol infusion decreases human cortical gamma-aminobutyric acid and N-acetylaspartate as measured with proton magnetic resonance spectroscopy at 4 tesla. Biol Psychiatry. 2012 Feb 1;71(3):239-46. doi: 10.1016/j.biopsych.2011.06.026. Epub 2011 Aug 19. PMID 21855054
- [Background] Grandjean EM, Berthet P, Ruffmann R, Leuenberger P. Efficacy of oral long-term N-acetylcysteine in chronic bronchopulmonary disease: a meta-analysis of published double-blind, placebo-controlled clinical trials. Clin Ther. 2000 Feb;22(2):209-21. doi: 10.1016/S0149-2918(00)88479-9. PMID 10743980
- [Background] Grant BF, Stinson FS, Dawson DA, Chou SP, Dufour MC, Compton W, Pickering RP, Kaplan K. Prevalence and co-occurrence of substance use disorders and independent mood and anxiety disorders: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Arch Gen Psychiatry. 2004 Aug;61(8):807-16. doi: 10.1001/archpsyc.61.8.807. PMID 15289279
- [Background] Grant JE, Odlaug BL, Chamberlain SR, Potenza MN, Schreiber LR, Donahue CB, Kim SW. A randomized, placebo-controlled trial of N-acetylcysteine plus imaginal desensitization for nicotine-dependent pathological gamblers. J Clin Psychiatry. 2014 Jan;75(1):39-45. doi: 10.4088/JCP.13m08411. PMID 24345329
- [Background] Grant JE, Odlaug BL, Kim SW. A double-blind, placebo-controlled study of N-acetyl cysteine plus naltrexone for methamphetamine dependence. Eur Neuropsychopharmacol. 2010 Nov;20(11):823-8. doi: 10.1016/j.euroneuro.2010.06.018. Epub 2010 Jul 22. PMID 20655182
- [Background] Gray KM, Carpenter MJ, Baker NL, DeSantis SM, Kryway E, Hartwell KJ, McRae-Clark AL, Brady KT. A double-blind randomized controlled trial of N-acetylcysteine in cannabis-dependent adolescents. Am J Psychiatry. 2012 Aug;169(8):805-12. doi: 10.1176/appi.ajp.2012.12010055. PMID 22706327
- [Background] Hafeman DM, Chang KD, Garrett AS, Sanders EM, Phillips ML. Effects of medication on neuroimaging findings in bipolar disorder: an updated review. Bipolar Disord. 2012 Jun;14(4):375-410. doi: 10.1111/j.1399-5618.2012.01023.x. PMID 22631621
- [Background] Hahn T, Dresler T, Ehlis AC, Plichta MM, Heinzel S, Polak T, Lesch KP, Breuer F, Jakob PM, Fallgatter AJ. Neural response to reward anticipation is modulated by Gray's impulsivity. Neuroimage. 2009 Jul 15;46(4):1148-53. doi: 10.1016/j.neuroimage.2009.03.038. Epub 2009 Mar 25. PMID 19328237
- [Background] Harris AD, Puts NA, Edden RA. Tissue correction for GABA-edited MRS: Considerations of voxel composition, tissue segmentation, and tissue relaxations. J Magn Reson Imaging. 2015 Nov;42(5):1431-40. doi: 10.1002/jmri.24903. Epub 2015 Jul 14. PMID 26172043
- [Background] Hassel S, Almeida JR, Kerr N, Nau S, Ladouceur CD, Fissell K, Kupfer DJ, Phillips ML. Elevated striatal and decreased dorsolateral prefrontal cortical activity in response to emotional stimuli in euthymic bipolar disorder: no associations with psychotropic medication load. Bipolar Disord. 2008 Dec;10(8):916-27. doi: 10.1111/j.1399-5618.2008.00641.x. PMID 19594507
- [Background] Hermann D, Weber-Fahr W, Sartorius A, Hoerst M, Frischknecht U, Tunc-Skarka N, Perreau-Lenz S, Hansson AC, Krumm B, Kiefer F, Spanagel R, Mann K, Ende G, Sommer WH. Translational magnetic resonance spectroscopy reveals excessive central glutamate levels during alcohol withdrawal in humans and rats. Biol Psychiatry. 2012 Jun 1;71(11):1015-21. doi: 10.1016/j.biopsych.2011.07.034. Epub 2011 Sep 10. PMID 21907974
- [Background] Hoblyn JC, Balt SL, Woodard SA, Brooks JO 3rd. Substance use disorders as risk factors for psychiatric hospitalization in bipolar disorder. Psychiatr Serv. 2009 Jan;60(1):50-5. doi: 10.1176/ps.2009.60.1.50. PMID 19114570
- [Background] Hoerst M, Weber-Fahr W, Tunc-Skarka N, Ruf M, Bohus M, Schmahl C, Ende G. Correlation of glutamate levels in the anterior cingulate cortex with self-reported impulsivity in patients with borderline personality disorder and healthy controls. Arch Gen Psychiatry. 2010 Sep;67(9):946-54. doi: 10.1001/archgenpsychiatry.2010.93. Epub 2010 Jul 5. PMID 20603446
- [Background] Holdiness MR. Clinical pharmacokinetics of N-acetylcysteine. Clin Pharmacokinet. 1991 Feb;20(2):123-34. doi: 10.2165/00003088-199120020-00004. PMID 2029805
- [Background] Horiuchi Y, Nakayama J, Ishiguro H, Ohtsuki T, Detera-Wadleigh SD, Toyota T, Yamada K, Nankai M, Shibuya H, Yoshikawa T, Arinami T. Possible association between a haplotype of the GABA-A receptor alpha 1 subunit gene (GABRA1) and mood disorders. Biol Psychiatry. 2004 Jan 1;55(1):40-5. doi: 10.1016/s0006-3223(03)00689-9. PMID 14706423
- [Background] Jones AL, Jarvie DR, Simpson D, Hayes PC, Prescott LF. Pharmacokinetics of N-acetylcysteine are altered in patients with chronic liver disease. Aliment Pharmacol Ther. 1997 Aug;11(4):787-91. doi: 10.1046/j.1365-2036.1997.00209.x. PMID 9305490
- [Background] Juenke JM, Wienhoff KA, Anderson BL, McMillin GA, Johnson-Davis KL. Performance characteristics of the ARK diagnostics gabapentin immunoassay. Ther Drug Monit. 2011 Aug;33(4):398-401. doi: 10.1097/FTD.0b013e318220bb65. PMID 21654348
- [Background] Kaladjian A, Jeanningros R, Azorin JM, Nazarian B, Roth M, Mazzola-Pomietto P. Reduced brain activation in euthymic bipolar patients during response inhibition: an event-related fMRI study. Psychiatry Res. 2009 Jul 15;173(1):45-51. doi: 10.1016/j.pscychresns.2008.08.003. Epub 2009 May 12. PMID 19442494
- [Background] Kalivas PW. The glutamate homeostasis hypothesis of addiction. Nat Rev Neurosci. 2009 Aug;10(8):561-72. doi: 10.1038/nrn2515. Epub 2009 Jul 1. PMID 19571793
- [Background] Kalivas PW, O'Brien C. Drug addiction as a pathology of staged neuroplasticity. Neuropsychopharmacology. 2008 Jan;33(1):166-80. doi: 10.1038/sj.npp.1301564. Epub 2007 Sep 5. PMID 17805308
- [Background] Kaufman RE, Ostacher MJ, Marks EH, Simon NM, Sachs GS, Jensen JE, Renshaw PF, Pollack MH. Brain GABA levels in patients with bipolar disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Apr 30;33(3):427-34. doi: 10.1016/j.pnpbp.2008.12.025. Epub 2009 Jan 10. PMID 19171176
- [Background] Knackstedt LA, LaRowe S, Mardikian P, Malcolm R, Upadhyaya H, Hedden S, Markou A, Kalivas PW. The role of cystine-glutamate exchange in nicotine dependence in rats and humans. Biol Psychiatry. 2009 May 15;65(10):841-5. doi: 10.1016/j.biopsych.2008.10.040. Epub 2008 Dec 21. PMID 19103434
- [Background] Koob GF, Volkow ND. Neurocircuitry of addiction. Neuropsychopharmacology. 2010 Jan;35(1):217-38. doi: 10.1038/npp.2009.110. PMID 19710631
- [Background] Krystal JH, Staley J, Mason G, Petrakis IL, Kaufman J, Harris RA, Gelernter J, Lappalainen J. Gamma-aminobutyric acid type A receptors and alcoholism: intoxication, dependence, vulnerability, and treatment. Arch Gen Psychiatry. 2006 Sep;63(9):957-68. doi: 10.1001/archpsyc.63.9.957. PMID 16952998
- [Background] Kuzniecky R, Ho S, Pan J, Martin R, Gilliam F, Faught E, Hetherington H. Modulation of cerebral GABA by topiramate, lamotrigine, and gabapentin in healthy adults. Neurology. 2002 Feb 12;58(3):368-72. doi: 10.1212/wnl.58.3.368. PMID 11839834
- [Background] LaRowe SD, Kalivas PW, Nicholas JS, Randall PK, Mardikian PN, Malcolm RJ. A double-blind placebo-controlled trial of N-acetylcysteine in the treatment of cocaine dependence. Am J Addict. 2013 Sep-Oct;22(5):443-52. doi: 10.1111/j.1521-0391.2013.12034.x. Epub 2013 May 15. PMID 23952889
- [Background] LaRowe SD, Myrick H, Hedden S, Mardikian P, Saladin M, McRae A, Brady K, Kalivas PW, Malcolm R. Is cocaine desire reduced by N-acetylcysteine? Am J Psychiatry. 2007 Jul;164(7):1115-7. doi: 10.1176/ajp.2007.164.7.1115. PMID 17606664
- [Background] Lawrence NS, Williams AM, Surguladze S, Giampietro V, Brammer MJ, Andrew C, Frangou S, Ecker C, Phillips ML. Subcortical and ventral prefrontal cortical neural responses to facial expressions distinguish patients with bipolar disorder and major depression. Biol Psychiatry. 2004 Mar 15;55(6):578-87. doi: 10.1016/j.biopsych.2003.11.017. PMID 15013826
- [Background] Le-Niculescu H, Patel SD, Bhat M, Kuczenski R, Faraone SV, Tsuang MT, McMahon FJ, Schork NJ, Nurnberger JI Jr, Niculescu AB 3rd. Convergent functional genomics of genome-wide association data for bipolar disorder: comprehensive identification of candidate genes, pathways and mechanisms. Am J Med Genet B Neuropsychiatr Genet. 2009 Mar 5;150B(2):155-81. doi: 10.1002/ajmg.b.30887. PMID 19025758
- [Background] Li CS, Luo X, Yan P, Bergquist K, Sinha R. Altered impulse control in alcohol dependence: neural measures of stop signal performance. Alcohol Clin Exp Res. 2009 Apr;33(4):740-50. doi: 10.1111/j.1530-0277.2008.00891.x. Epub 2009 Jan 21. PMID 19170662
- [Background] Luijten M, Machielsen MW, Veltman DJ, Hester R, de Haan L, Franken IH. Systematic review of ERP and fMRI studies investigating inhibitory control and error processing in people with substance dependence and behavioural addictions. J Psychiatry Neurosci. 2014 May;39(3):149-69. doi: 10.1503/jpn.130052. PMID 24359877
- [Background] MacKinnon DP, Fairchild AJ, Fritz MS. Mediation analysis. Annu Rev Psychol. 2007;58:593-614. doi: 10.1146/annurev.psych.58.110405.085542. PMID 16968208
- [Background] Madayag A, Lobner D, Kau KS, Mantsch JR, Abdulhameed O, Hearing M, Grier MD, Baker DA. Repeated N-acetylcysteine administration alters plasticity-dependent effects of cocaine. J Neurosci. 2007 Dec 19;27(51):13968-76. doi: 10.1523/JNEUROSCI.2808-07.2007. PMID 18094234
- [Background] Maeng S, Zarate CA Jr, Du J, Schloesser RJ, McCammon J, Chen G, Manji HK. Cellular mechanisms underlying the antidepressant effects of ketamine: role of alpha-amino-3-hydroxy-5-methylisoxazole-4-propionic acid receptors. Biol Psychiatry. 2008 Feb 15;63(4):349-52. doi: 10.1016/j.biopsych.2007.05.028. Epub 2007 Jul 23. PMID 17643398
- [Background] Mason BJ, Quello S, Goodell V, Shadan F, Kyle M, Begovic A. Gabapentin treatment for alcohol dependence: a randomized clinical trial. JAMA Intern Med. 2014 Jan;174(1):70-7. doi: 10.1001/jamainternmed.2013.11950. PMID 24190578
- [Background] Mason GF, Petrakis IL, de Graaf RA, Gueorguieva R, Guidone E, Coric V, Epperson CN, Rothman DL, Krystal JH. Cortical gamma-aminobutyric acid levels and the recovery from ethanol dependence: preliminary evidence of modification by cigarette smoking. Biol Psychiatry. 2006 Jan 1;59(1):85-93. doi: 10.1016/j.biopsych.2005.06.009. Epub 2005 Nov 14. PMID 16289397
- [Background] Massat I, Souery D, Del-Favero J, Oruc L, Noethen MM, Blackwood D, Thomson M, Muir W, Papadimitriou GN, Dikeos DG, Kaneva R, Serretti A, Lilli R, Smeraldi E, Jakovljevic M, Folnegovic V, Rietschel M, Milanova V, Valente F, Van Broeckhoven C, Mendlewicz J. Excess of allele1 for alpha3 subunit GABA receptor gene (GABRA3) in bipolar patients: a multicentric association study. Mol Psychiatry. 2002;7(2):201-7. doi: 10.1038/sj.mp.4000953. PMID 11840313
- [Background] McFarland K, Kalivas PW. The circuitry mediating cocaine-induced reinstatement of drug-seeking behavior. J Neurosci. 2001 Nov 1;21(21):8655-63. doi: 10.1523/JNEUROSCI.21-21-08655.2001. PMID 11606653
- [Background] Michael N, Erfurth A, Ohrmann P, Gossling M, Arolt V, Heindel W, Pfleiderer B. Acute mania is accompanied by elevated glutamate/glutamine levels within the left dorsolateral prefrontal cortex. Psychopharmacology (Berl). 2003 Jul;168(3):344-6. doi: 10.1007/s00213-003-1440-z. Epub 2003 Apr 9. PMID 12684737
- [Background] Michael N, Erfurth A, Pfleiderer B. Elevated metabolites within dorsolateral prefrontal cortex in rapid cycling bipolar disorder. Psychiatry Res. 2009 Apr 30;172(1):78-81. doi: 10.1016/j.pscychresns.2009.01.002. Epub 2009 Feb 23. PMID 19239983
- [Background] Mitchell JM, Fields HL, D'Esposito M, Boettiger CA. Impulsive responding in alcoholics. Alcohol Clin Exp Res. 2005 Dec;29(12):2158-69. doi: 10.1097/01.alc.0000191755.63639.4a. PMID 16385186
- [Background] Mon A, Durazzo TC, Meyerhoff DJ. Glutamate, GABA, and other cortical metabolite concentrations during early abstinence from alcohol and their associations with neurocognitive changes. Drug Alcohol Depend. 2012 Sep 1;125(1-2):27-36. doi: 10.1016/j.drugalcdep.2012.03.012. Epub 2012 Apr 12. PMID 22503310
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Mousavi SG, Sharbafchi MR, Salehi M, Peykanpour M, Karimian Sichani N, Maracy M. The efficacy of N-acetylcysteine in the treatment of methamphetamine dependence: a double-blind controlled, crossover study. Arch Iran Med. 2015 Jan;18(1):28-33. PMID 25556383
- [Background] Mullins PG, Chen H, Xu J, Caprihan A, Gasparovic C. Comparative reliability of proton spectroscopy techniques designed to improve detection of J-coupled metabolites. Magn Reson Med. 2008 Oct;60(4):964-9. doi: 10.1002/mrm.21696. PMID 18816817
- [Background] Murphy ER, Fernando AB, Urcelay GP, Robinson ES, Mar AC, Theobald DE, Dalley JW, Robbins TW. Impulsive behaviour induced by both NMDA receptor antagonism and GABAA receptor activation in rat ventromedial prefrontal cortex. Psychopharmacology (Berl). 2012 Jan;219(2):401-10. doi: 10.1007/s00213-011-2572-1. Epub 2011 Nov 19. PMID 22101355
- [Background] Myrick H, Anton RF, Li X, Henderson S, Drobes D, Voronin K, George MS. Differential brain activity in alcoholics and social drinkers to alcohol cues: relationship to craving. Neuropsychopharmacology. 2004 Feb;29(2):393-402. doi: 10.1038/sj.npp.1300295. PMID 14679386
- [Background] Myrick H, Anton RF, Li X, Henderson S, Randall PK, Voronin K. Effect of naltrexone and ondansetron on alcohol cue-induced activation of the ventral striatum in alcohol-dependent people. Arch Gen Psychiatry. 2008 Apr;65(4):466-75. doi: 10.1001/archpsyc.65.4.466. PMID 18391135
- [Background] Myrick H, Li X, Randall PK, Henderson S, Voronin K, Anton RF. The effect of aripiprazole on cue-induced brain activation and drinking parameters in alcoholics. J Clin Psychopharmacol. 2010 Aug;30(4):365-72. doi: 10.1097/JCP.0b013e3181e75cff. PMID 20571434
- [Background] Myrick H, Malcolm R, Randall PK, Boyle E, Anton RF, Becker HC, Randall CL. A double-blind trial of gabapentin versus lorazepam in the treatment of alcohol withdrawal. Alcohol Clin Exp Res. 2009 Sep;33(9):1582-8. doi: 10.1111/j.1530-0277.2009.00986.x. Epub 2009 May 26. PMID 19485969
- [Background] Murali AR, Attar BM, Katz A, Kotwal V, Clarke PM. Utility of Platelet Count for Predicting Cirrhosis in Alcoholic Liver Disease: Model for Identifying Cirrhosis in a US Population. J Gen Intern Med. 2015 Aug;30(8):1112-7. doi: 10.1007/s11606-015-3238-1. Epub 2015 Feb 21. PMID 25701049
- [Background] Nery FG, Stanley JA, Chen HH, Hatch JP, Nicoletti MA, Monkul ES, Lafer B, Soares JC. Bipolar disorder comorbid with alcoholism: a 1H magnetic resonance spectroscopy study. J Psychiatr Res. 2010 Apr;44(5):278-85. doi: 10.1016/j.jpsychires.2009.09.006. Epub 2009 Oct 8. PMID 19818454
- [Background] Niciu MJ, Luckenbaugh DA, Ionescu DF, Richards EM, Vande Voort JL, Ballard ED, Brutsche NE, Furey ML, Zarate CA Jr. Riluzole likely lacks antidepressant efficacy in ketamine non-responders. J Psychiatr Res. 2014 Nov;58:197-9. doi: 10.1016/j.jpsychires.2014.07.022. Epub 2014 Aug 6. No abstract available. PMID 25139008
- [Background] Ogg RJ, Zou P, Allen DN, Hutchins SB, Dutkiewicz RM, Mulhern RK. Neural correlates of a clinical continuous performance test. Magn Reson Imaging. 2008 May;26(4):504-12. doi: 10.1016/j.mri.2007.09.004. Epub 2008 Feb 20. PMID 18068933
- [Background] O'Gorman RL, Michels L, Edden RA, Murdoch JB, Martin E. In vivo detection of GABA and glutamate with MEGA-PRESS: reproducibility and gender effects. J Magn Reson Imaging. 2011 May;33(5):1262-7. doi: 10.1002/jmri.22520. PMID 21509888
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Ongur D, Jensen JE, Prescot AP, Stork C, Lundy M, Cohen BM, Renshaw PF. Abnormal glutamatergic neurotransmission and neuronal-glial interactions in acute mania. Biol Psychiatry. 2008 Oct 15;64(8):718-726. doi: 10.1016/j.biopsych.2008.05.014. Epub 2008 Jul 7. PMID 18602089
- [Background] Oquendo MA, Currier D, Liu SM, Hasin DS, Grant BF, Blanco C. Increased risk for suicidal behavior in comorbid bipolar disorder and alcohol use disorders: results from the National Epidemiologic Survey on Alcohol and Related Conditions (NESARC). J Clin Psychiatry. 2010 Jul;71(7):902-9. doi: 10.4088/JCP.09m05198gry. PMID 20667292
- [Background] Otani K, Ujike H, Tanaka Y, Morita Y, Katsu T, Nomura A, Uchida N, Hamamura T, Fujiwara Y, Kuroda S. The GABA type A receptor alpha5 subunit gene is associated with bipolar I disorder. Neurosci Lett. 2005 Jun 10-17;381(1-2):108-13. doi: 10.1016/j.neulet.2005.02.010. Epub 2005 Feb 25. PMID 15882799
- [Background] Pattij T, Vanderschuren LJ. The neuropharmacology of impulsive behaviour. Trends Pharmacol Sci. 2008 Apr;29(4):192-9. doi: 10.1016/j.tips.2008.01.002. Epub 2008 Mar 4. PMID 18304658
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Peng PW, Wijeysundera DN, Li CC. Use of gabapentin for perioperative pain control -- a meta-analysis. Pain Res Manag. 2007 Summer;12(2):85-92. doi: 10.1155/2007/840572. PMID 17505569
- [Background] Perlis RH, Dennehy EB, Miklowitz DJ, Delbello MP, Ostacher M, Calabrese JR, Ametrano RM, Wisniewski SR, Bowden CL, Thase ME, Nierenberg AA, Sachs G. Retrospective age at onset of bipolar disorder and outcome during two-year follow-up: results from the STEP-BD study. Bipolar Disord. 2009 Jun;11(4):391-400. doi: 10.1111/j.1399-5618.2009.00686.x. PMID 19500092
- [Background] Petroff OA, Hyder F, Rothman DL, Mattson RH. Effects of gabapentin on brain GABA, homocarnosine, and pyrrolidinone in epilepsy patients. Epilepsia. 2000 Jun;41(6):675-80. doi: 10.1111/j.1528-1157.2000.tb00227.x. PMID 10840398
- [Background] Petroff OA, Rothman DL, Behar KL, Lamoureux D, Mattson RH. The effect of gabapentin on brain gamma-aminobutyric acid in patients with epilepsy. Ann Neurol. 1996 Jan;39(1):95-9. doi: 10.1002/ana.410390114. PMID 8572673
- [Background] Petty F, Kramer GL, Dunnam D, Rush AJ. Plasma GABA in mood disorders. Psychopharmacol Bull. 1990;26(2):157-61. PMID 2236451
- [Background] Phan KL, Fitzgerald DA, Cortese BM, Seraji-Bozorgzad N, Tancer ME, Moore GJ. Anterior cingulate neurochemistry in social anxiety disorder: 1H-MRS at 4 Tesla. Neuroreport. 2005 Feb 8;16(2):183-6. doi: 10.1097/00001756-200502080-00024. PMID 15671874
- [Background] Phillips ML, Travis MJ, Fagiolini A, Kupfer DJ. Medication effects in neuroimaging studies of bipolar disorder. Am J Psychiatry. 2008 Mar;165(3):313-20. doi: 10.1176/appi.ajp.2007.07071066. Epub 2008 Feb 1. PMID 18245175
- [Background] Post RM, Denicoff KD, Leverich GS, Altshuler LL, Frye MA, Suppes TM, Rush AJ, Keck PE Jr, McElroy SL, Luckenbaugh DA, Pollio C, Kupka R, Nolen WA. Morbidity in 258 bipolar outpatients followed for 1 year with daily prospective ratings on the NIMH life chart method. J Clin Psychiatry. 2003 Jun;64(6):680-90; quiz 738-9. doi: 10.4088/jcp.v64n0610. PMID 12823083
- [Background] Prado E, Maes M, Piccoli LG, Baracat M, Barbosa DS, Franco O, Dodd S, Berk M, Vargas Nunes SO. N-acetylcysteine for therapy-resistant tobacco use disorder: a pilot study. Redox Rep. 2015 Sep;20(5):215-22. doi: 10.1179/1351000215Y.0000000004. Epub 2015 Mar 2. PMID 25729878
- [Background] Prescot AP, Locatelli AE, Renshaw PF, Yurgelun-Todd DA. Neurochemical alterations in adolescent chronic marijuana smokers: a proton MRS study. Neuroimage. 2011 Jul 1;57(1):69-75. doi: 10.1016/j.neuroimage.2011.02.044. Epub 2011 Feb 22. PMID 21349338
- [Background] Prescot AP, Renshaw PF, Yurgelun-Todd DA. gamma-Amino butyric acid and glutamate abnormalities in adolescent chronic marijuana smokers. Drug Alcohol Depend. 2013 May 1;129(3):232-9. doi: 10.1016/j.drugalcdep.2013.02.028. Epub 2013 Mar 21. PMID 23522493
- [Background] Prescot AP, Renshaw PF. Two-dimensional J-resolved proton MR spectroscopy and prior knowledge fitting (ProFit) in the frontal and parietal lobes of healthy volunteers: assessment of metabolite discrimination and general reproducibility. J Magn Reson Imaging. 2013 Mar;37(3):642-51. doi: 10.1002/jmri.23848. Epub 2012 Oct 10. PMID 23055387
- [Background] Prisciandaro JJ, Brown DG, Brady KT, Tolliver BK. Comorbid anxiety disorders and baseline medication regimens predict clinical outcomes in individuals with co-occurring bipolar disorder and alcohol dependence: Results of a randomized controlled trial. Psychiatry Res. 2011 Aug 15;188(3):361-5. doi: 10.1016/j.psychres.2011.04.030. Epub 2011 Jun 8. PMID 21641663
- [Background] Prisciandaro JJ, DeSantis SM, Chiuzan C, Brown DG, Brady KT, Tolliver BK. Impact of depressive symptoms on future alcohol use in patients with co-occurring bipolar disorder and alcohol dependence: a prospective analysis in an 8-week randomized controlled trial of acamprosate. Alcohol Clin Exp Res. 2012 Mar;36(3):490-6. doi: 10.1111/j.1530-0277.2011.01645.x. Epub 2011 Sep 20. PMID 21933201
- [Background] Prisciandaro JJ, Joseph JE, Myrick H, McRae-Clark AL, Henderson S, Pfeifer J, Brady KT. The relationship between years of cocaine use and brain activation to cocaine and response inhibition cues. Addiction. 2014 Dec;109(12):2062-70. doi: 10.1111/add.12666. Epub 2014 Jul 21. PMID 24938849
- [Background] Prisciandaro JJ, Myrick H, Henderson S, McRae-Clark AL, Brady KT. Prospective associations between brain activation to cocaine and no-go cues and cocaine relapse. Drug Alcohol Depend. 2013 Jul 1;131(1-2):44-9. doi: 10.1016/j.drugalcdep.2013.04.008. Epub 2013 May 15. PMID 23683790
- [Background] Prisciandaro JJ, Rembold J, Brown DG, Brady KT, Tolliver BK. Predictors of clinical trial dropout in individuals with co-occurring bipolar disorder and alcohol dependence. Drug Alcohol Depend. 2011 Nov 1;118(2-3):493-6. doi: 10.1016/j.drugalcdep.2011.03.029. Epub 2011 May 6. PMID 21549529
- [Background] Prisciandaro JJ, Schacht JP, Prescot AP, Renshaw PF, Brown TR, Anton RF. Associations Between Recent Heavy Drinking and Dorsal Anterior Cingulate N-Acetylaspartate and Glutamate Concentrations in Non-Treatment-Seeking Individuals with Alcohol Dependence. Alcohol Clin Exp Res. 2016 Mar;40(3):491-6. doi: 10.1111/acer.12977. Epub 2016 Feb 8. PMID 26853538
- [Background] Prisciandaro JJ, Tolliver BK. Evidence for the continuous latent structure of mania and depression in out-patients with bipolar disorder: results from the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). Psychol Med. 2015;45(12):2595-603. doi: 10.1017/S0033291715000513. Epub 2015 Apr 17. PMID 25881582
- [Background] Provencher SW. Estimation of metabolite concentrations from localized in vivo proton NMR spectra. Magn Reson Med. 1993 Dec;30(6):672-9. doi: 10.1002/mrm.1910300604. PMID 8139448
- [Background] Puts NA, Edden RA. In vivo magnetic resonance spectroscopy of GABA: a methodological review. Prog Nucl Magn Reson Spectrosc. 2012 Jan;60:29-41. doi: 10.1016/j.pnmrs.2011.06.001. Epub 2011 Jun 12. No abstract available. PMID 22293397
- [Background] Regier DA, Farmer ME, Rae DS, Locke BZ, Keith SJ, Judd LL, Goodwin FK. Comorbidity of mental disorders with alcohol and other drug abuse. Results from the Epidemiologic Catchment Area (ECA) Study. JAMA. 1990 Nov 21;264(19):2511-8. PMID 2232018
- [Background] Robinson ES, Eagle DM, Economidou D, Theobald DE, Mar AC, Murphy ER, Robbins TW, Dalley JW. Behavioural characterisation of high impulsivity on the 5-choice serial reaction time task: specific deficits in 'waiting' versus 'stopping'. Behav Brain Res. 2009 Jan 23;196(2):310-6. doi: 10.1016/j.bbr.2008.09.021. Epub 2008 Oct 2. PMID 18940201
- [Background] Rose MA, Kam PC. Gabapentin: pharmacology and its use in pain management. Anaesthesia. 2002 May;57(5):451-62. doi: 10.1046/j.0003-2409.2001.02399.x. PMID 11966555
- [Background] Rosner S, Hackl-Herrwerth A, Leucht S, Lehert P, Vecchi S, Soyka M. Acamprosate for alcohol dependence. Cochrane Database Syst Rev. 2010 Sep 8;2010(9):CD004332. doi: 10.1002/14651858.CD004332.pub2. PMID 20824837
- [Background] Rowland LM, Bustillo JR, Mullins PG, Jung RE, Lenroot R, Landgraf E, Barrow R, Yeo R, Lauriello J, Brooks WM. Effects of ketamine on anterior cingulate glutamate metabolism in healthy humans: a 4-T proton MRS study. Am J Psychiatry. 2005 Feb;162(2):394-6. doi: 10.1176/appi.ajp.162.2.394. PMID 15677610
- [Background] Rubio G, Jimenez M, Rodriguez-Jimenez R, Martinez I, Avila C, Ferre F, Jimenez-Arriero MA, Ponce G, Palomo T. The role of behavioral impulsivity in the development of alcohol dependence: a 4-year follow-up study. Alcohol Clin Exp Res. 2008 Sep;32(9):1681-7. doi: 10.1111/j.1530-0277.2008.00746.x. Epub 2008 Jul 9. PMID 18631324
- [Background] Salloum IM, Cornelius JR, Daley DC, Kirisci L, Himmelhoch JM, Thase ME. Efficacy of valproate maintenance in patients with bipolar disorder and alcoholism: a double-blind placebo-controlled study. Arch Gen Psychiatry. 2005 Jan;62(1):37-45. doi: 10.1001/archpsyc.62.1.37. PMID 15630071
- [Background] Sanacora G, Zarate CA, Krystal JH, Manji HK. Targeting the glutamatergic system to develop novel, improved therapeutics for mood disorders. Nat Rev Drug Discov. 2008 May;7(5):426-37. doi: 10.1038/nrd2462. PMID 18425072
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Schacht JP, Anton RF, Myrick H. Functional neuroimaging studies of alcohol cue reactivity: a quantitative meta-analysis and systematic review. Addict Biol. 2013 Jan;18(1):121-33. doi: 10.1111/j.1369-1600.2012.00464.x. Epub 2012 May 10. PMID 22574861
- [Background] Schacht JP, Anton RF, Randall PK, Li X, Henderson S, Myrick H. Stability of fMRI striatal response to alcohol cues: a hierarchical linear modeling approach. Neuroimage. 2011 May 1;56(1):61-8. doi: 10.1016/j.neuroimage.2011.02.004. Epub 2011 Feb 18. PMID 21316465
- [Background] Schmaal L, Veltman DJ, Nederveen A, van den Brink W, Goudriaan AE. N-acetylcysteine normalizes glutamate levels in cocaine-dependent patients: a randomized crossover magnetic resonance spectroscopy study. Neuropsychopharmacology. 2012 Aug;37(9):2143-52. doi: 10.1038/npp.2012.66. Epub 2012 May 2. PMID 22549117
- [Background] Schulte RF, Boesiger P. ProFit: two-dimensional prior-knowledge fitting of J-resolved spectra. NMR Biomed. 2006 Apr;19(2):255-63. doi: 10.1002/nbm.1026. PMID 16541464
- [Background] Sills GJ. The mechanisms of action of gabapentin and pregabalin. Curr Opin Pharmacol. 2006 Feb;6(1):108-13. doi: 10.1016/j.coph.2005.11.003. Epub 2005 Dec 22. PMID 16376147
- [Background] Silveri MM, Sneider JT, Crowley DJ, Covell MJ, Acharya D, Rosso IM, Jensen JE. Frontal lobe gamma-aminobutyric acid levels during adolescence: associations with impulsivity and response inhibition. Biol Psychiatry. 2013 Aug 15;74(4):296-304. doi: 10.1016/j.biopsych.2013.01.033. Epub 2013 Mar 14. PMID 23498139
- [Background] Simon JJ, Walther S, Fiebach CJ, Friederich HC, Stippich C, Weisbrod M, Kaiser S. Neural reward processing is modulated by approach- and avoidance-related personality traits. Neuroimage. 2010 Jan 15;49(2):1868-74. doi: 10.1016/j.neuroimage.2009.09.016. Epub 2009 Sep 18. PMID 19770056
- [Background] Simon NM, Otto MW, Wisniewski SR, Fossey M, Sagduyu K, Frank E, Sachs GS, Nierenberg AA, Thase ME, Pollack MH. Anxiety disorder comorbidity in bipolar disorder patients: data from the first 500 participants in the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD). Am J Psychiatry. 2004 Dec;161(12):2222-9. doi: 10.1176/appi.ajp.161.12.2222. PMID 15569893
- [Background] Smith SM, Jenkinson M, Woolrich MW, Beckmann CF, Behrens TE, Johansen-Berg H, Bannister PR, De Luca M, Drobnjak I, Flitney DE, Niazy RK, Saunders J, Vickers J, Zhang Y, De Stefano N, Brady JM, Matthews PM. Advances in functional and structural MR image analysis and implementation as FSL. Neuroimage. 2004;23 Suppl 1:S208-19. doi: 10.1016/j.neuroimage.2004.07.051. PMID 15501092
- [Background] Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend. 1996 Sep;42(1):49-54. doi: 10.1016/0376-8716(96)01263-x. PMID 8889403
- [Background] Soeiro-de-Souza MG, Henning A, Machado-Vieira R, Moreno RA, Pastorello BF, da Costa Leite C, Vallada H, Otaduy MC. Anterior cingulate Glutamate-Glutamine cycle metabolites are altered in euthymic bipolar I disorder. Eur Neuropsychopharmacol. 2015 Dec;25(12):2221-9. doi: 10.1016/j.euroneuro.2015.09.020. Epub 2015 Oct 9. PMID 26476706
- [Background] Soeiro-de-Souza MG, Salvadore G, Moreno RA, Otaduy MC, Chaim KT, Gattaz WF, Zarate CA Jr, Machado-Vieira R. Bcl-2 rs956572 polymorphism is associated with increased anterior cingulate cortical glutamate in euthymic bipolar I disorder. Neuropsychopharmacology. 2013 Feb;38(3):468-75. doi: 10.1038/npp.2012.203. Epub 2012 Oct 17. PMID 23072837
- [Background] Stone JM, Dietrich C, Edden R, Mehta MA, De Simoni S, Reed LJ, Krystal JH, Nutt D, Barker GJ. Ketamine effects on brain GABA and glutamate levels with 1H-MRS: relationship to ketamine-induced psychopathology. Mol Psychiatry. 2012 Jul;17(7):664-5. doi: 10.1038/mp.2011.171. Epub 2012 Jan 3. No abstract available. PMID 22212598
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Swann AC. The strong relationship between bipolar and substance-use disorder. Ann N Y Acad Sci. 2010 Feb;1187:276-93. doi: 10.1111/j.1749-6632.2009.05146.x. PMID 20201858
- [Background] Swann AC, Lijffijt M, Lane SD, Steinberg JL, Moeller FG. Increased trait-like impulsivity and course of illness in bipolar disorder. Bipolar Disord. 2009 May;11(3):280-8. doi: 10.1111/j.1399-5618.2009.00678.x. PMID 19419385
- [Background] Swann AC, Lijffijt M, Lane SD, Steinberg JL, Moeller FG. Severity of bipolar disorder is associated with impairment of response inhibition. J Affect Disord. 2009 Jul;116(1-2):30-6. doi: 10.1016/j.jad.2008.10.022. Epub 2008 Nov 26. PMID 19038460
- [Background] Swann AC, Pazzaglia P, Nicholls A, Dougherty DM, Moeller FG. Impulsivity and phase of illness in bipolar disorder. J Affect Disord. 2003 Jan;73(1-2):105-11. doi: 10.1016/s0165-0327(02)00328-2. PMID 12507743
- [Background] Swick D, Ashley V, Turken U. Are the neural correlates of stopping and not going identical? Quantitative meta-analysis of two response inhibition tasks. Neuroimage. 2011 Jun 1;56(3):1655-65. doi: 10.1016/j.neuroimage.2011.02.070. Epub 2011 Mar 3. PMID 21376819
- [Background] Thoma R, Mullins P, Ruhl D, Monnig M, Yeo RA, Caprihan A, Bogenschutz M, Lysne P, Tonigan S, Kalyanam R, Gasparovic C. Perturbation of the glutamate-glutamine system in alcohol dependence and remission. Neuropsychopharmacology. 2011 Jun;36(7):1359-65. doi: 10.1038/npp.2011.20. Epub 2011 Mar 9. PMID 21389979
- [Background] Tolliver BK, Desantis SM, Brown DG, Prisciandaro JJ, Brady KT. A randomized, double-blind, placebo-controlled clinical trial of acamprosate in alcohol-dependent individuals with bipolar disorder: a preliminary report. Bipolar Disord. 2012 Feb;14(1):54-63. doi: 10.1111/j.1399-5618.2011.00973.x. PMID 22329472
- [Background] Umhau JC, Momenan R, Schwandt ML, Singley E, Lifshitz M, Doty L, Adams LJ, Vengeliene V, Spanagel R, Zhang Y, Shen J, George DT, Hommer D, Heilig M. Effect of acamprosate on magnetic resonance spectroscopy measures of central glutamate in detoxified alcohol-dependent individuals: a randomized controlled experimental medicine study. Arch Gen Psychiatry. 2010 Oct;67(10):1069-77. doi: 10.1001/archgenpsychiatry.2010.125. PMID 20921123
- [Background] van Veenendaal TM, IJff DM, Aldenkamp AP, Hofman PA, Vlooswijk MC, Rouhl RP, de Louw AJ, Backes WH, Jansen JF. Metabolic and functional MR biomarkers of antiepileptic drug effectiveness: A review. Neurosci Biobehav Rev. 2015 Dec;59:92-9. doi: 10.1016/j.neubiorev.2015.10.004. Epub 2015 Oct 22. PMID 26475992
- [Background] Wang PW, Sailasuta N, Chandler RA, Ketter TA. Magnetic resonance spectroscopic measurement of cerebral gamma-aminobutyric acid concentrations in patients with bipolar disorders. Acta Neuropsychiatr. 2006 Apr;18(2):120-6. doi: 10.1111/j.1601-5215.2006.00132.x. PMID 26989801
- [Background] Wilk J, West JC, Rae DS, Regier DA. Relationship of comorbid substance and alcohol use disorders to disability among patients in routine psychiatric practice. Am J Addict. 2006 Mar-Apr;15(2):180-5. doi: 10.1080/10550490500528799. PMID 16595357
- [Background] Wrase J, Schlagenhauf F, Kienast T, Wustenberg T, Bermpohl F, Kahnt T, Beck A, Strohle A, Juckel G, Knutson B, Heinz A. Dysfunction of reward processing correlates with alcohol craving in detoxified alcoholics. Neuroimage. 2007 Apr 1;35(2):787-94. doi: 10.1016/j.neuroimage.2006.11.043. Epub 2007 Feb 8. PMID 17291784
- [Background] Yoon YH, Chen CM, Yi HY, Moss HB. Effect of comorbid alcohol and drug use disorders on premature death among unipolar and bipolar disorder decedents in the United States, 1999 to 2006. Compr Psychiatry. 2011 Sep-Oct;52(5):453-64. doi: 10.1016/j.comppsych.2010.10.005. Epub 2010 Dec 13. PMID 21146814
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Yuksel C, Ongur D. Magnetic resonance spectroscopy studies of glutamate-related abnormalities in mood disorders. Biol Psychiatry. 2010 Nov 1;68(9):785-94. doi: 10.1016/j.biopsych.2010.06.016. Epub 2010 Aug 21. PMID 20728076
- [Background] Zand L, McKian KP, Qian Q. Gabapentin toxicity in patients with chronic kidney disease: a preventable cause of morbidity. Am J Med. 2010 Apr;123(4):367-73. doi: 10.1016/j.amjmed.2009.09.030. PMID 20362757

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin, Washout, Then N-Acetylcysteine, Washout, Then Placebo Oral Capsule, Washout: Three, 1-week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
- N-Acetylcysteine, Washout, Then Placebo Oral Capsule, Washout, Then Gabapentin, Washout: 3, 1 week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
- Placebo Oral Tablet, Washout, Then Gabapentin, Washout, Then N-Acetylcysteine, Washout: Three, 1-week conditions. Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
- Placebo Oral Capsule, Washout, Then N-Acetylcysteine, Washout, Then Gabapentin, Washout: Three, 1-week conditions. Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
- Gabapentin, Washout, Then Placebo Oral Capsule, Washout, Then N-Acetylcysteine, Washout: Three, 1-week conditions. Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
- N-Acetylcysteine, Washout, Then Gabapentin, Washout, Then Placebo Oral Capsule, Washout: Three, 1-week conditions. Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg Week 3 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
Period: Overall Study
Arm/Group | Gabapentin, Washout, Then N-Acetylcysteine, Washout, Then Placebo Oral Capsule, Washout | N-Acetylcysteine, Washout, Then Placebo Oral Capsule, Washout, Then Gabapentin, Washout | Placebo Oral Tablet, Washout, Then Gabapentin, Washout, Then N-Acetylcysteine, Washout | Placebo Oral Capsule, Washout, Then N-Acetylcysteine, Washout, Then Gabapentin, Washout | Gabapentin, Washout, Then Placebo Oral Capsule, Washout, Then N-Acetylcysteine, Washout | N-Acetylcysteine, Washout, Then Gabapentin, Washout, Then Placebo Oral Capsule, Washout
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed | 7 | 8 | 8 | 5 | 8 | 7
Not Completed | 2 | 1 | 1 | 4 | 1 | 2
Not completed — Claustrophobia | 0 | 1 | 1 | 0 | 1 | 0
Not completed — MRI Equipment Failure | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Inclimate Weather | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Potential presence of non-MRI safe metal in body | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin, Then N-Acetylcysteine, Then Placebo Oral Capsule | N-Acetylcysteine, Then Placebo Oral Capsule, Then Gabapentin | Placebo Oral Tablet, Then Gabapentin, Then N-Acetylcysteine | Placebo Oral Capsule, Then N-Acetylcysteine, Then Gabapentin | Gabapentin, Then Placebo Oral Capsule, Then N-Acetylcysteine | N-Acetylcysteine, Then Gabapentin, Then Placebo Oral Capsule | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 9 | 9 | 54
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 41.33 [21 to 60] | 41.22 [24 to 61] | 41.11 [24 to 61] | 39.44 [20 to 50] | 42.44 [20 to 62] | 38.22 [22 to 57] | 40.63 [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 5 | 6 | 5 | 31
  Male | 4 | 4 | 4 | 4 | 3 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 9 | 9 | 9 | 9 | 7 | 9 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 2 | 3 | 2 | 1 | 13
  White | 6 | 6 | 7 | 6 | 6 | 8 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 9 | 9 | 54

OUTCOME MEASURES:

1. Primary Outcome: Prefrontal GABA+ Concentrations
Description: Concentrations of GABA+, referenced to unsuppressed water and corrected for within-voxel CSF proportion, in dorsal anterior cingulate cortex measured via Proton Magnetic Resonance Spectroscopy (i.e., MEGA-PRESS).
Time Frame: Day 5 of each experimental condition
Population: Overall number of participants analyzed includes participants who completed the entire medication condition (i.e. participants who started N-Acetylcysteine, Gabapentin, or Placebo Oral Tablet but who did not complete the MRI portion of the condition have been removed from outcome measure data analysis, but are included in other portions of this study record [Adverse Events, Demographics, etc.]).
Measure: Mean (Standard Deviation); unit: mmol/kg
Groups:
- N-Acetylcysteine: Each 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 2,400mg N-acetylcysteine) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  N-Acetylcysteine: 5 day trial of N-acetylcysteine with titration to 2,400mg
- Gabapentin: Each 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
- Placebo Oral Tablet: Each 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Tablet: 5 day trial of matched placebo
Arm/Group | N-Acetylcysteine | Gabapentin | Placebo Oral Tablet
Number analyzed (Participants) | 43 | 41 | 46
mmol/kg | 3.90 (0.543) | 3.93 (0.646) | 3.73 (0.705)

2. Primary Outcome: Prefrontal Glx Concentrations
Description: Concentrations of Glx (i.e., glutamate + glutamine), referenced to unsuppressed water and corrected for within-voxel CSF proportion, in dorsal anterior cingulate cortex measured via Proton Magnetic Resonance Spectroscopy.
Time Frame: Day 5 of each experimental condition
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/kg
Arm/Group | N-Acetylcysteine | Gabapentin | Placebo Oral Tablet
Number analyzed (Participants) | 43 | 41 | 46
mmol/kg | 21.59 (2.518) | 21.69 (2.499) | 22.25 (2.746)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected over each participant's total study duration. This duration was a 3-week period for each participant (i.e. 3, 1-week condition periods). Adverse event data collection took place for the entirety of the study which was 6 years.
Description: At each study visit following the initial screening visit, study participants were assessed by the study medical doctor for any adverse events. Adverse events were recorded, rated on a severity scale, determined their relation to the study medication, and any treatment or intervention needed was discussed. The study medical doctor followed up with all previously reported adverse events at the following visits to determine if the events had ceased.
Arm/Group | N-Acetylcysteine | Gabapentin | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 10/48 | 9/48 | 6/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=48) | Gabapentin (N=48) | Placebo Oral Tablet (N=51)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Memory Impairment (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mood Swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dissociation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Teeth Grinding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin Odor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT03220776/Prot_SAP_000.pdf